CLINICAL TRIAL: NCT02398045
Title: Developing Computerised Cognitive Behavioural Therapy for Adults With Obsessive-compulsive Disorder
Brief Title: Developing Computerised CBT for Adults With OCD
Acronym: CCBT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry, London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David Veale, Dr, Institute of Psychiatry, London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCBT-1111; 658-PAHTLZB (Other Grant/Funding Number: Maudsley Charity)
Record Dates: First submitted 2014-06-04; First posted 2015-03-25 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-02

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; cognitive behavioural therapy; computerised
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computerised CBT (Experimental): Computerised CBT for OCD
  Interventions: Other: Computerised CBT for OCD

INTERVENTIONS:
Other: Computerised CBT for OCD — Computerised CBT for OCD

SUMMARY:
The study aims to pilot a new computerised cognitive behavioural therapy programme for a small case series of adults with obsessive-compulsive disorder. The investigators hypothesise that the findings will demonstrate improvements in symptomatology following the programme. The programme will have longer-term aims of being rolled out over a number of IAPT services within the NHS, reducing waiting lists and increasing therapist time.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over with OCD as defined by DSM-IV who are seeking CBT.
* The patient describes their OCD as their main problem and scores between 14 and 30 on the YBOCS (Goodman et al, 1989). A score above 30 is in the severe range and indicates that the CBT should probably be therapist delivered.
* Able to use self-help materials in English and answer written questionnaires.
* Able to access the internet (either at home or in a public library or drop in centre or at the clinic).
* Have a current episode of OCD of more than 6 months in duration.

Exclusion Criteria:

* Significant and complex co-morbidity (e.g. significant personality disorder, severe depression or alcohol dependence, which requires longer therapy or is more difficult to treat). Such patients are likely to be part of a Community Mental Health team or be funded by the Department of Health's National Specialist Commissioning Team scheme for severe treatment refectory OCD.
* Current active suicidal intent or severe self-neglect that requires hospitalisation.
* The patient has a primary problem of compulsive hoarding (as such patients are more complex or are more likely to be under a Community Mental Health team).
* Continuing to receive another form of psychotherapy.
* Has received CBT for OCD in the past year.
* A participant may be taking an anti-depressant for OCD but must be on a stable dose for at least 12 weeks prior to entry in the trial with no plans to alter the dose during the trial period. There must also be no plan to commence on an anti-depressant or anti-psychotic medication. (Participants excluded because of their current or planned medication may be offered a further assessment for the trial after being on a stable dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Y-BOCS-OCD | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
  Yale-Brown Obsessive-Compulsive Scale for OCD. Questions focus on obsessive thoughts participants may have along with behaviours they feel compelled to do in order to reduce their anxiety. This outcome is expected to change (improve) from baseline throughout the trial as a result of the computerised CBT.

SECONDARY OUTCOMES:
Psychiatric Diagnostic Screening Questionnaire | baseline
  This form asks participants about emotions, mood, thoughts, and behaviours and asks patients to describe how they've been acting, feeling or thinking. Questions refer specifically to either the last 2 weeks or the last 6 months (and specify which when necessary).
DSM-IV OCD SCID | baseline
  This is used to check that participants meet the DSM-IV diagnosis for Obsessive-Compulsive Disorder and covers a range of questions from any previous treatment received to alcohol and drug consumption.
Patient Health Questionnaire | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
Generalised anxiety disorder assessment | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
  This is a 7 item scale asking about anxiety levels over the past 2 weeks.
Work and social adjustment scale | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
  This scale has 5 questions, each of which is answered using a 9 point likert scale. It focuses on work, home management, social and private leisure activities, and relationships/family.
Expectation for treatment success and credibility | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
  Based on the information collected from all other measures, a therapist or clinician will make a prediction about the participants suitability for treatment using CBT, and how well (or not well) they expect the participant to respond to CBT treatment.
demographic variables | baseline
  This involves questions about Age, gender, ethnicity, education, employment, relationship status and access to the internet.
Obsessive-compulsive inventory | baseline, week 3, week 4 or week 5 after baseline, 12 weeks, 1 month follow-up
  This measure involved 42 statements relating to distress that people may experience in their everyday lives. Participants will answer each statement on a likert scale from 0-4 in terms of how much that experience has bothered them during the past month.

CONTACTS AND LOCATIONS:
Overall Officials: David Veale, MRCPsych, Principal Investigator — Institute of Psychiatry
Locations (2):
- United Kingdom (2):
  - Centre for Anxiety Disorders and Trauma, London, London
  - South London and Maudsley NHS Trust, London